CLINICAL TRIAL: NCT00299247
Title: SP Resistance Markers and Falciparum Malaria Transmission
Brief Title: SP Resistance and Falciparum Malaria Transmission
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-246
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2010-01

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria, Plasmodium falciparum, drug resistance, Colombia
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: sulfadoxine/pyrimethamine

SUMMARY:
The purpose of this study is to study resistance to current malaria treatments and affordable alternatives for uncomplicated malaria. Resistance occurs in areas where these treatments are used frequently. This study may help prevent future resistance. About 150 residents in Buenaventura, Colombia will participate. They will have uncomplicated malaria and they will be followed for 28 days after treatment. Physical exams and blood draws are included in study visits.

DETAILED DESCRIPTION:
Drug-resistant Plasmodium falciparum is a major threat to global public health and new strategies are needed to deter spread of resistance to available and forthcoming antimalarial drugs. This study seeks to contribute to understanding the molecular basis of spread of drug resistance in a setting with low level of sulfadoxine-pyrimethamine (SP) treatment failure. The objectives of this study are to compare the prevalence of dihydrofolate reductase (DHFR) and dihydropteroate synthase (DHPS) point mutations associated with SP resistance before and after SP treatment of uncomplicated Plasmodium falciparum malaria episodes and to measure parasite infectivity to Anopheles mosquitoes of post-treatment gametocytes with and without DHFR and DHPR mutations. Patients with uncomplicated falciparum malaria will receive a standard SP regimen and will be closely followed for 28 days. This study will add new knowledge of the understanding of ways in which resistance is spread and is expected to provide a sound basis for the future clinical evaluation of antimalarial drug combinations designed to prevent transmission of drug-resistance malaria.

ELIGIBILITY:
Inclusion Criteria:

Age more than 5 years Positive blood smear for falciparum malaria Informed consent from participant or parent Intention to remain in the study area for at least 4 weeks from the time of enrollment

Exclusion Criteria:

Mixed Plasmodium infection Parasitemia > 10% Hematocrit < 15% Respiratory distress Spontaneous bleeding (from gums, nose, gastrointestinal tract, etc.) Recent seizures or coma Prostration or weakness, so that the patient cannot sit or walk, with no obvious neurological explanation Inability to drink Persistent vomiting History of allergy or adverse reaction to sulfadoxine-pyrimethamine (SP) or sulfa drugs Known pregnancy

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2006-12 (Estimated); Study Completion 2006-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Malaria Vaccine and Drug Development Center, Cali
  - Universidad del Valle Sede San Fernando, Cali